CLINICAL TRIAL: NCT04226456
Title: Clinical Trial: Intratympanic Injection of N-acetylcysteine for Protection of Cisplatin-induced Ototoxicity
Brief Title: Intratympanic Administration of N-acetylcysteine for Protection of Cisplatin-induced Ototoxicity
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUB-NAC
Record Dates: First submitted 2019-12-09; First posted 2020-01-13 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-02

CONDITIONS: Ototoxic Hearing Loss; Ototoxic Hearing Loss, Bilateral; Ototoxicity; Tinnitus
MeSH Terms: conditions — Ototoxicity; Tinnitus | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Standard arm (Arm A): Cisplatin from 70 to 100 mg/m2 intravenous (IV) once for 3 to 7 cycles +/- Radiotherapy (depending on the type and the severity of the neoplastic disease)
  Dosis and number of Cisplatin cycles are determined by the oncologist depending on type and severity of neoplastic disease.
- N-acetylcysteine (Experimental): Experimental arm (Arm B):
  * 0.4 to 1 ml of NAC 10% through intratympanic injection (ITI) from 40 to 60 minutes maximum prior to each Cisplatin cycle.
  * Cisplatin from 70 to 100 mg/m2 intravenous (IV) once for 3 to 7 cycles +/- Radiotherapy (depending on the type and the severity of the neoplastic disease)
  Dosis and number of Cisplatin cycles are determined by the oncologist depending on type and severity of neoplastic disease.
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine — Injection of a 10% solution of N-acetylcysteine through transtympanic injection in both ears
  Other Names: Lysomucil 10%
  Arms: N-acetylcysteine

SUMMARY:
The purpose of this study is to assess the efficacity of N-acetylcystein against Cisplatin-induced ototoxicity.

DETAILED DESCRIPTION:
This is a monocentric, randomized, controlled, open label phase IV superiority trial.

After signing the informed consent form and upon the confirmation of the patient eligibility, patients will be randomized 1:1 to the experimental arm (NAC + Cisplatin) or the standard arm (Cisplatin).

The primary objective of this trial is to evaluate the protecting effect of Lysomucil® 10% against Cisplatin-induced ototoxicity. In this case, we will evaluate its effect through the transtympanic administration in both ears.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18-year-old
* Patients suffering from a neoplastic disease for which treatment protocol includes Cisplatin.

Exclusion Criteria:

* Women of childbearing potential pregnant or with intention to become pregnant within the trial duration
* Women who are breastfeeding
* Pathological findings on otoscopy that do not allow safe intratympanic drug delivery.
* Conductive hearing loss > 20dBHL
* Meniere disease
* Medical history of sudden hearing loss
* Sensoryneural Hearing loss (SNHL) with mean ≥ 40dbHL Pure Tonal Audiometry (PTA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Apparition of ototoxicity | 6 month after last injection
  the apparition of ototoxicity as defined by the International Common Terminology Criteria for Adverse Events (CTCAE), version 5:
  * A Threshold shift of 15 - 25 decibel (dB) averaged at 2 contiguous test frequencies in at least one ear
  * and/or the apparition of a tinnitus (not previously present).

SECONDARY OUTCOMES:
Evaluate the apparition of ototoxicity defined by the inclusion of high frequency audiometry (Tune Grading System) | 6 month after last injection
  the apparition of ototoxicity as defined by the International Common Terminology Criteria for Adverse Events (CTCAE), version 5:
  * A Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear
  * and/or the apparition of a tinnitus (not previously present).
Hearing quality of life: Evaluation of the Impact of Hearing Loss in Adults ERSA | 6 month after last injection
  Evaluation of the Impact of Hearing Loss in Adults (ERSA) For each question, the score of 0 means maximal difficulties, the sore of 10 means ideal situation Formulation is uniform, with no inversions: 0 always corresponds to maximal difficulty and 10 to an ideal situation, so that the lower the score the greater the impact of hearing loss on quality of life. Maximum score is 200 for respondents in work and 150 for those not in work or in retirement.
Hearing quality of life: Tinnitus Handicap Index (THI) | 6 month after last injection
  Tinnitus Handicap Index (THI) score Range : 0 to 100. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan Cavelier, MD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- CHU Saint-Pierre, Brussels, Belgium